CLINICAL TRIAL: NCT04438980
Title: Treatment of COVID-19 Pneumonia With Glucocorticoids. A Randomized Controlled Trial
Brief Title: Glucocorticoids in COVID-19 (CORTIVID)
Acronym: CORTIVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Complejo Hospitalario de Navarra (Other); Hospital Sant Joan Despí Moisès Broggi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORTIVID
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Covid-19 Pneumonia
Keywords: Covid-19; pneumonia; Inflammatory phase; Glucocorticoids
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone Arm (Experimental): Standard of care plus Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Placebo Arm (Placebo Comparator): Standard of care plus placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — -A dose of 120 mg/day of methylprednisolone for 3 days, administered by intravenous infusión
  Arms: Methylprednisolone Arm
Other: Placebo — -An infusion bag of 100 mL of 0.9% saline
  Arms: Placebo Arm

SUMMARY:
Around 30% of admitted patients with COVID-19 pneumonia develop a hyper-inflammatory state whose progression to an acute respiratory distress syndrome (ARSD) could be prevented by the early initiation of immune-modulatory agents. The role of glucocorticoids (GC) in this setting remains controversial. This study aims to assess the safety and effectiveness of GC pulses to improve the clinical outcomes of patients with COVID-19 pneumonia with risen inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Diagnosis of SARS-CoV-2 pneumonia confirmed by reverse transcriptase polymerase chain reaction (RT-PCR) on nasopharyngeal swab or sputum according to the recommendations of the Spanish Ministry of Health.
* Length of symptoms consistent with COVID-19 ≥7 days.
* Hospital admission.
* At least one of the following: CRP >60 mg/L, IL-6 >40 pg/mL, ferritin >1000 μg/L.
* Acceptation of informed consent

Exclusion Criteria:

* Allergy or contraindication to any of the drugs under study.
* SpO2 <90% (in air ambient) or PaO2 <60 mmHg (in ambient air) or PaO2/FiO2 <300 mmHg.
* Ongoing treatment with glucocorticoids, immunosuppressive, or biologic drugs with another indication.
* Decompensated diabetes mellitus.
* Uncontrolled hypertension.
* Psychotic or manic disorder.
* Active cancer.
* Pregnancy or lactation.
* Clinical or biochemical suspicion (procalcitonin >0.5 ng/mL) of active infection other than SARS-CoV-2.
* Out-of-hospital management patient.
* Conservative or palliative management patient.
* Participation in another clinical trial.
* Any important and uncontrolled medical, psychological, psychiatric, geographic or social problem that contraindicates the patient's participation in the trial or that does not allow adequate follow-up and adherence to the protocol and evaluation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing treatment failure | At 14 days after randomization
  • Death
Proportion of patients developing treatment failure | At 14 days after randomization
  • Need for admission in an intensive care unit (ICU)
Proportion of patients developing treatment failure | At 14 days after randomization
  • Need for mechanical ventilation
Proportion of patients developing treatment failure | At 14 days after randomization
  • Decrease in SpO2 <90% (in ambient air) or PaO2 <60 mmHg (in ambient air) or PaO2FiO2 <300 mmHg, associated with radiological impairment

SECONDARY OUTCOMES:
Mortality at day 28 | At 28 days after randomization
Proportion of patients requiring ICU admission | At 28 days after randomization
Proportion of patients requiring rescue-therapy with tocilizumab | At 14 days after randomization
Length of hospital stay | At 28 days after randomization
  Time in days from randomization until the date of hospital discharge.
Proportion of severe adverse events | At 28 days after randomization
  Any undesirable experience related to the use of the studied drugs, which causes patient's death, life-threatening risk, hospitalization or extension of a previous hospitalization, disability or permanent damage, requires intervention to prevent permanent impairment or damage, or is considered medically relevant
Proportion of bacterial, fungal or opportunistic infections | At 28 days after randomization
Evolution of inflammatory biomarkers related to COVID-19 | At 14 days after randomization
  Change in plasma levels of C-reactive protein (CRP)
Evolution of inflammatory biomarkers related to COVID-19 | At 14 days after randomization
  Change in plasma levels of ferritin
Evolution of inflammatory biomarkers related to COVID-19 | At 14 days after randomization
  Change in plasma levels of interleukin-6 (IL-6)
Evolution of inflammatory biomarkers related to COVID-19 | At 14 days after randomization
  Change in plasma levels of lactate dehydrogenase (LDH)
Evolution of inflammatory biomarkers related to COVID-19 | At 14 days after randomization
  Change in plasma levels of D-dimer (DD)
Proportion of SARS-CoV-2 clearance. | At 7 days after randomization
  Negativization of RT-PCR for SARS-CoV-2 on nasopharyngeal swab or sputum

CONTACTS AND LOCATIONS:
Overall Officials: Iñigo Les Bujanda, PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (2):
- Spain (2):
  - Hospital Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be available for exploitation in future research projects. This statement also includes the availability of the study protocol, the statistical analysis plan, the informed consent form, the clinical study report and the analytic code.

REFERENCES:
- [Derived] Les Bujanda I, Loureiro-Amigo J, Bastons FC, Guerra IE, Sanchez JA, Murgadella-Sancho A, Rey RG, Lopez JL, Alvarez JS. Treatment of COVID-19 pneumonia with glucocorticoids (CORTIVID): a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Jan 11;22(1):43. doi: 10.1186/s13063-020-04999-4. PMID 33430891